CLINICAL TRIAL: NCT00154752
Title: A Randomized Trial Comparing Concurrent Chemoradiation Versus Wide Pelvic Lymphadenectomy for Advanced Rectal Cancer
Brief Title: Concurrent Chemoradiation Versus Wide Pelvic Lymphadenectomy for Advanced Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9100013841
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-11-22 (Estimated); Status verified 1999-01

CONDITIONS: Colorectal Cancer
Keywords: Rectal cancer, CCRT, Pelvic lymphadenoectomy.
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

INTERVENTIONS:
Procedure: CCRT, Pelvic lymphadenoectomy.

SUMMARY:
Based on the neurophysiology, it is well known that sympathetic nerves control the ejaculatory function and bladder neck closure. In contrast, the parasympathetic nerves control penile erection and bladder wall contraction. Because of the difference in cultural background of the patients and training background of the physicians between Western and Oriental Countries, the Western people did not believe in the efficacy of wide pelvic lymphadenectomy. In the Oriental countries, due to the shortage of standardized facilities, treatment protocol, and manpower, the concurrent preoperative chemoradiation therapy (CCRT) of American style is currently not widely accepted. Therefore, the advantage and disadvantage of these two treatment modalities for advanced rectal cancers need be further clarified. In this project, we plan to randomly assign the patients into two groups: (1) concurrent preoperative chemoradiation therapy (CCRT) + conventional surgery group; (2) wide pelvic lymphadenectomy group. Thereafter, we plan to evaluate: (1) the anorectal function by anorectal manometry and colonic transit time using radioopaque markers; (2) the micturition function using urodynamic study; (3) the penile erection by RigiScan; and (4) the ejaculatory function by clinical interview of the patients. Moreover, the various clinicopathologic factors, including the depth of tumor invasion and the status of lymph node invasion, were recorded in detail according to the guidelines recommended by the Japanese Society of Coloproctology. Furthermore, we will evaluate the oncological results for these patients.

DETAILED DESCRIPTION:
This project is in continuation of our previous study (NTUH92-S044) and is focused on the comparison of the advantage and disadvantage of the following two treatment modalities: (1) preoperative neoadjuvant therapy (CCRT) followed by conventional surgery; (2) the Japanese-style of wide pelvic lymphadenectomy, for the treatment of potentially operable locally advanced rectal cancer. It is well-known that the keypoint for the surgical treatment of rectal cancer is to achieve a balance between 'radical resection of the tumor' and 'functional preservation for the pelvic organs'. Primary adenocarcinoma of the rectum is generally characterized by localized and comparatively slow-growing, as compared to the fast-growing tumors of other gastrointestinal malignancies. Thus, extended systemic pelvic lymphadenectomy has been considered the best choice for cure. However, there is major difference of concept between the Western and Oriental colorectal surgeons regarding the appropriate extent of lymphadenectomy for the treatment of rectal cancers lying below the peritoneal reflection. Theoretically, there are two major pathways for the lymphatic drainage of lower rectal cancers: one is upward to the root of inferior mesenteric artery (IMA); the other is along the middle hemorrhoidal artery to the obturator fossa. Because the American people tend to be very fatty and the pelvic lymphadenectomy is difficult to perform, most rectal cancer patients receive conventional limited resection combined with aggressive chemotherapy and pelvic irradiation. In contrast, because the Oriental people are thinner and pelvic lymphadenectomy is easier to perform, and most important of all, the Japanese surgeons were very meticulous in cancer surgery, the extended pelvic lymphadenectomy has become the routine procedure for the advanced lower rectal cancer in Japan. However, extended pelvic lymphadenectomy can inevitably cause the autonomic nerve damage, which thereafter result in the disturbance of micturition and sexual function. To overcome this genitourinary complication, the Japanese surgeon developed the autonomic nerve-sparing surgery. Generally speaking, pelvic autonomic nerves consist of sympathetic signals via the paired hypogastric nerves and paired sacral splanchnic nerves, and the parasympathetic signals via the pelvic splanchnic nerves. The sympathetic and parasympathetic fibers intermingled with each other to form the pelvic plexus, which is located at the lateral side of the lateral ligament. Pelvic plexus then send the composite autonomic signals to innervate distal rectum and genitourinary organs. Thus, the injury of autonomic nerve can reflect the functional disorder of the anorectum and genitourinary organs. Based on the neurophysiology, it is well known that sympathetic nerves control the ejaculatory function and bladder neck closure. In contrast, the parasympathetic nerves control penile erection and bladder wall contraction. Because of the difference in cultural background of the patients and training background of the physicians between Western and Oriental Countries, the Western people did not believe in the efficacy of wide pelvic lymphadenectomy. In the Oriental countries, due to the shortage of standardized facilities, treatment protocol, and manpower, the concurrent preoperative chemoradiation therapy (CCRT) of American style is currently not widely accepted. Therefore, the advantage and disadvantage of these two treatment modalities for advanced rectal cancers need be further clarified. In this project, we plan to randomly assign the patients into two groups: (1) concurrent preoperative chemoradiation therapy (CCRT) + conventional surgery group; (2) wide pelvic lymphadenectomy group. Thereafter, we plan to evaluate: (1) the anorectal function by anorectal manometry and colonic transit time using radioopaque markers; (2) the micturition function using urodynamic study ; (3) the penile erection by RigiScan; and (4) the ejaculatory function by clinical interview of the patients. Moreover, the various clinicopathologic factors, including the depth of tumor invasion and the status of lymph node invasion, were recorded in detail according to the guidelines recommended by the Japanese Society of Coloproctology. Furthermore, we will evaluate the oncological results for these patients. There are 2 characteristics for this project: (1) This is a randomized, prospective study which has not been conducted in the literature; (2) The functional evaluation is conducted in an objective way which is different from the reported series based only on the subjective patient interview.

During the conduction of our precious project (NTU 92-S044), we found that the response rate of locally advanced rectal cancer after CCRT is satisfactory. The response rate is even more increased after the addition of oxaliplatin to the traditional regimen of 5-Fu plus leucovorin. However, there was no significance patients between these 2 allocated groups of patients in terms of genitourinary dysfunction. These preliminary data need be further testified by accrual of more patients with longer time of follow-up. Therefore, it is mandatory for us to further perform this project. We believe that this study will provide a new balance point between the 'radical resection' and the 'functional preservation' for advanced rectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary rectal adenocarcinoma below the peritoneal reflection 2. Tumor with suspected lateral nodes involvement and/or T4 lesion 3. ASA class Ⅰto Ⅲ patients 4. The life expectancy was greater than 12 weeks 5. Age of the patients between 18 and 75 years

Exclusion Criteria:

* 1. Emergency operation 2. Primary tumors with distant metastasis or peritoneal carcinomatosis 3. Primary tumors located at other anatomical sites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1999-01; Study Completion 2005-06

PRIMARY OUTCOMES:
oncologic results

SECONDARY OUTCOMES:
functional results

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung Liang, M.D., Ph.D., Principal Investigator — Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C.
Locations (1):
- Department of Surgery, National Taiwan University Hospital, No.7, Chung-Shan South Road, Taipei, TAIWAN, R.O.C., Taipei, Taiwan